CLINICAL TRIAL: NCT00055926
Title: A Phase I Safety and Pharmacokinetic/Pharmacodynamic Study of CP-724, 714 In Patients With Metastatic HER2-Overexpressing Breast Cancer
Brief Title: CP-724,714 in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000271533; UCLA-0209105; PFIZER-A4031001
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — 2-methoxy-N-(3-(4-((3-methyl-4-((6-methyl-3-pyridinyl)oxy)phenyl)amino)-6-quinazolinyl)-2-propenyl)acetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CP-724,714

SUMMARY:
RATIONALE: CP-724,714 may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth.

PURPOSE: Phase I trial to study the effectiveness of CP-724,714 in treating patients who have metastatic HER2-overexpressing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of CP-724,714 in patients with metastatic HER2-overexpressing breast cancer.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine, preliminarily, any antitumor activity of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the relationship of drug-related adverse events to pharmacokinetic exposure parameters in these patients.
* Determine the relationship of changes in serum HER2 extracellular domain and HER2 receptor tyrosine kinase phosphorylation to pharmacokinetic exposure parameters and clinical outcome in patients treated with this drug.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive oral CP-724,714 on days 1 and 3-21 during course 1 and then daily during subsequent courses. Courses repeat every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of CP-724,714 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for at least 30 days.

PROJECTED ACCRUAL: A total of 3-20 patients will be accrued for this study within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2-overexpressing breast cancer
* Prior or newly documented HER2 amplification by fluorescence in situ hybridization (FISH)
* Progressive metastatic disease
* Must have received at least one prior chemotherapy regimen for metastatic breast cancer
* At least 1 measurable or evaluable lesion
* At least 1 lesion accessible for 2 separate core biopsies for pharmacodynamic evaluation
* 18 and over
* Male or female
* ECOG 0-1
* Life expectancy, More than 3 months
* Hematopoietic

  * Absolute neutrophil count at least 1,500/mm^3*
  * Platelet count at least 100,000/mm^3* NOTE: *Without hematopoietic growth factors or transfusions
* Hepatic

  * Bilirubin no greater than 1.5 mg/dL
  * AST/ALT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Renal

  * Creatinine no greater than 1.5 times ULN OR
  * Creatinine clearance at least 60 mL/min
* Cardiovascular

  * 12-lead ECG with normal tracing
* history of cardiovascular disease (i.e., ischemic heart disease, arrhythmia, or congestive heart failure) unless asymptomatic for the past year with no requirement for antiarrhythmics or a clinically significant medical management change
* Gastrointestinal

  * Able to take oral medication* Negative pregnancy test
  * Fertile patients must use effective contraception
* At least 4 weeks since prior trastuzumab (Herceptin)
* At least 4 weeks since other prior biologic therapy or immunotherapy
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)
* At least 6 months since prior doxorubicin or doxorubicin equivalents without any prior or developing signs or symptoms of cardiomyopathy
* No cumulative doses of more than 300 mg/m^2
* At least 2 weeks since prior hormonal therapy for the primary disease
* Concurrent hormone replacement therapy or luteinizing hormone-releasing hormone agonists allowed
* At least 4 weeks since prior radiotherapy
* At least 3 weeks since prior major surgery (2 weeks for minor surgery)
* Recovered from prior therapy
* At least 4 weeks since prior investigational treatment
* Coumarin or heparin derivatives allowed for the prevention of deep vein thrombosis or port patency

Exclusion Criteria:

* known or clinically suspected brain metastases or leptomeningeal disease
* symptomatic edema or third-space fluid (e.g., ascites or pleural effusions)
* known hepatitis B or C infection
* significant ECG changes that require medical intervention
* QTc interval less than 460 msec
* No history of torsade or other symptomatic QTc abnormality
* LVEF greater than 50% by MUGA
* gastrointestinal abnormality that would require medications (including all antacids)
* persistent symptoms of an esophageal or digestive disorder
* pregnant or nursing
* known HIV infection
* active infection
* concurrent uncontrolled systemic disorders or laboratory abnormalities that would preclude study drug safety evaluation
* mental disorder that would preclude study compliance or ability to give informed consent
* No more than 2 prior trastuzumab-based regimens for advanced disease
* concurrent immunotherapy
* more than 1 prior anthracycline- or anthracenedione-containing regimen (except with approval of the sponsor)
* prior high-dose chemotherapy with hematopoietic stem cell transplantation
* concurrent anticancer chemotherapy
* No concurrent anticancer hormonal therapy, including tamoxifen
* prior radiotherapy to the only disease site that would be assessed for response
* concurrent radiotherapy
* prior partial or complete gastrectomy
* concurrent antiarrhythmics
* concurrent antacids
* concurrent anticoagulant at therapeutic doses
* other concurrent experimental anticancer medications for breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-01; Primary Completion 2004-12 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Britten, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States